CLINICAL TRIAL: NCT05572307
Title: Peripheral Blood Single Cell Sequencing Analysis of Postoperative Delirium (POD) and Chronic Postsurgical Pain (CPSP) in Elderly Patients After Total Knee Arthroplasty
Brief Title: Peripheral Blood Single Cell Sequencing Analysis of POD and CPSP in Elderly Patients After Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuzhou Central Hospital (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XuzhouCH20221010
Record Dates: First submitted 2022-09-29; First posted 2022-10-07 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Delirium; Chronic Postsurgical Pain
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nucleated cells from peripheral blood were extracted and frozen.These cells are destroyed after single-cell sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- POD group: According to the occurrence of postoperative delirium, the patients were divided into POD group and non-POD group
- non-POD group: According to the occurrence of postoperative delirium, the patients were divided into POD group and non-POD group
- CPSP group: Patients were divided into CPSP group and non-CPSP group according to the occurrence of postoperative chronic pain
- non-CSP group: Patients were divided into CPSP group and non-CPSP group according to the occurrence of postoperative chronic pain

SUMMARY:
Single-celled sequencing for evaluating differences in gene expression patterns in different cell types of the dynamics of a means of this research as a starting point, to study the postoperative delirium and chronic pain at the cellular level changes the contents of a cell, reveal its occurrence and development of the role of gene regulation, find targets and biomarkers, and to provide new ideas for its pathogenesis, To provide theoretical basis support for its prevention, clinical diagnosis and treatment.

DETAILED DESCRIPTION:
The aim of this study was to investigate leukocyte heterogeneity in patients undergoing total knee arthroplasty with POD, paired non-POD patients, and cognitively normal healthy subjects by single cell sequencing, and to investigate leukocyte heterogeneity in patients with chronic pain and patients with pain relief after surgery through postoperative pain follow-up. Moreover, multi-omics single cell technology is used to analyze various cellular contents in a single cell simultaneously, which can capture molecular footprints with higher resolution. Comprehensive analysis of multiple omics datasets reveals the relationships between cellular patterns, establishes complex regulatory networks, and provides a holistic view of cellular state. From a single cell level analysis of POD and occurred in patients with chronic pain in patients with the characteristics of the white blood cells, looking for the peripheral immune system in the pathogenesis of the POD and the potential role of chronic pain occurs, may provide POD pathogenesis and chronic pain occurred an important visual Angle, may also help to provide POD biomarkers and therapeutic targets, To provide a possible solution for the prevention and treatment of postoperative delirium and postoperative chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old, regardless of gender.
* total knee arthroplasty for the first time.
* The ASA classification is I-Ⅲ.

Exclusion Criteria:

* severe neurological or psychiatric disorders
* drug and alcohol abuse
* patients on antidepressants
* failure and decompensation of vital organs
* chronic pain from previous surgery or trauma

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients undergoing elective total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of single cell sequencing before and after surgery | 1 day before surgery，1 day after surgery
  Leukocytes were isolated from peripheral blood and then sorted for subsequent single-cell sequencing analysis. Unbiased, high-throughput and high-resolution transcriptome analysis of single cells can reveal the gene structure and gene expression status of single cells, reflect the heterogeneity between cells, classify and analyze them, and carry out personalized research
3-minute Diagnostic Interview for CAM (3D-CAM) | Consecutive 7 days after the surgery
  Postoperative delirium was assessed by 3-minute Diagnostic Interview for confusion assessment method (CAM).
Visual analogue scale（VAS） | 3 months after the surgery
  A moving scale measuring about 10cm in length was used, with 10 scales on one side and "0" and "10" ends, respectively, with 0 indicating no pain and 10 indicating the most severe pain that could not be endured.
Short form McGill pain questionnaire（SF-MPQ） | 3 months after the surgery
  SF-MPQ is composed of sensory and emotional descriptors of pain, current pain intensity and visual analogue scale.
Leeds Assessment of Neuropathic Symptoms and Signs（LANSS） | 3 months after the surgery
  Make the needle perpendicular to the patient's skin, and apply different pressure on the skin to determine whether the patient has touch-induced pain.
Pain catastrophizing scale(PCS) | 3 months after the surgery
  PCS is defined as a belief system, a coping strategy and an evaluation process when experiencing and feeling pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yangzi Zhu, Doctor, Principal Investigator — Xuzhou Central Hospital; Liwei Wang, Doctor, Study Director — Xuzhou Central Hospital; Junli Cao, Doctor, Study Director — Jiangsu Province Key Laboratory of Anesthesiology, Xuzhou Medical University; Daqing Ma, Doctor, Study Chair — Imperial College London, Chelsea and Westminster Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No